CLINICAL TRIAL: NCT04048837
Title: Prospective Study for the Evaluation of Dengue Prognostic Biomarkers in Singapore
Status: Completed | Type: Observational
Sponsor: National University Hospital, Singapore (Other)
Collaborators: Tan Tock Seng Hospital (Other); Ng Teng Fong General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PrognosDen
Record Dates: First submitted 2018-10-19; First posted 2019-08-07 (Actual); Last update posted 2019-09-13 (Actual); Status verified 2019-09

CONDITIONS: Dengue Hemorrhagic Fever; Dengue Shock Syndrome; Severe Dengue
Keywords: Dengue
MeSH Terms: conditions — Severe Dengue; Dengue

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma and serum sample will be stored if patient agreeable to keep for future research.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
World Health Organisation (WHO) has identified Dengue as the fastest spreading mosquito-borne disease in the world. This study follows on from the National Medical Research Council STOP Dengue Translational and Clinical Research flagship grant. Differential serum concentrations of alpha2-macroglobulin (A2M), chymase (CMA1) and vascular endothelial growth factor A (VEGFA) were discovered to accurately identify dengue patients who will develop severe disease from those who will not, prior to the development of severe complications. By identifying patients at risk of developing severe disease in advance, these patients can be monitored more closely to provide more timely fluid interventions, and hopefully further reduce fatality rate. At the same time, more patients who are not at risk can be managed as outpatients to further minimize unnecessary hospitalization costs and wastage of healthcare resources. After discovery of the Dengue prognostic biomarkers, a multivariate logistic regression predictive model was built from a small retrospective derivative cohort (50 subjects), followed by validation using a small prospective validation cohort (50 subjects). The model had a receiver operating characteristic (ROC) curve AUC (area under the curve) of 0.944, and a sensitivity and specificity of 90% and 91% during validation, respectively. The premise of this study is to validate our observations in a larger prospective cohort (200 subjects). At the same time, we would like to better understand the characteristics of the Dengue prognostic biomarkers, especially whether there are situations in which the biomarkers cannot predict Dengue Haemorrhagic Fever (DHF)/ Dengue Shock Syndrome (DSS) and/or Severe Dengue (SD) and how the biomarkers can further improve the cost-effectiveness of the clinical management of Dengue patients.

DETAILED DESCRIPTION:
This is a non-interventional, prospective study aim to recruit 200 subjects from National University Hospital, Tan Tock Seng Hospital and Ng Teng Feng General Hospital over a period of 2 years to determine whether differential serum A2M, CMA1 and VEGFA concentrations can predict whether a dengue patient will develop severe disease. Serum A2M, CMA1 and VEGFA concentrations will be quantitated using enzyme-linked immunosorbent assays. The objectives of this study as below:

1. Determine the optimum cut-off for the prediction of DHF/DSS (WHO 1997 classification) and Severe Dengue (SD; WHO 2009 classification).
2. Better understand the characteristics (e.g. daily kinetics) of A2M, CMA1 and VEGFA in Dengue and how their serum concentrations are affected by other variables e.g. patient age and gender, day of sample collection, primary/secondary infection (based on patient memory and/or Standard Diagnostics SD BIOLINE Dengue Duo) and virus serotype.
3. Perform a cost-effectiveness analysis for the adoption of such a Dengue prognostic technology in hospital.

Eligible participants will be aged 21 and above with a laboratory confirmed dengue patients (either positive PCR or positive NS1), and meet all inclusion/exclusion criteria. Each participant will be given an information sheet and informed consent obtained from him/her. Blood will be drawn for PCR Dengue serotyping and measurements of serum concentrations of A2M, CMA1 and VEGFA via quantitative enzyme-linked immunosorbent assays (ELISA). Blood collection will be performed on the day of recruitment.

Participants may be managed as inpatients or outpatients as decided by their treating physician. For participants who are managed as Dengue outpatients, they will be asked to return to the outpatient clinic every day. For both Dengue inpatient and outpatient participants, blood will be drawn every day until they are discharged from care or Day 7 of the study, whichever earlier. If the participants are discharged from care (discharge from hospital or dengue clinic) on the day of recruitment, they will be asked to come back for study visit on Day 2. And 2 ml of blood will be collected for research purpose on Day 2. On the day of discharge, for both Dengue inpatients and outpatients, participants will each be given a questionnaire to complete. A separate questionnaire will also be filled up by the study team for the discharge of each Dengue inpatient participant. Should the participant be discharged prior to Day 7 of the study, a telephone call will be made to the discharged participant on Day 7 of the study to establish his/her health status. Upon completion of the study, each participant will be reimbursed a lump sum of $50.

Data collected will be entered into a paper case report forms and will be transcribed onto eCRF. All participants identifiers will not be collected. The system will allow for audit tracking. During the course of the study, auditors from relevant authorities may visit the study site to review protocol compliance, check electronic case report form (eCRFs) and ensure that the study is being conducted according to Good Clinical Practice (GCP).

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed Dengue i.e. laboratory confirmation of acute Dengue for this current disease episode by either (i) Positive polymerase chain reaction (PCR) for viral ribonucleic acid (RNA), or (ii) Positive NS1 antigen test with a compatible clinical syndrome
2. At least 21 years of age based on his/her birthday, and
3. Willing and able to give informed consent.

Exclusion Criteria:

1. Already classified as having Dengue Haemorrhagic Fever or Dengue Shock Syndrome (WHO 1997 classification) or severe Dengue (WHO 2009 classification) when they first present themselves to the hospital.
2. Assessed by Investigators to be unlikely to comply with trial procedures.
3. Have known or suspected congenital or acquired immunodeficiency, immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the past 6 months or long term corticosteroid therapy.
4. Have received blood or blood-derived products in the past three months that might interfere with the assessment of the biomarker responses.
5. Have participated in another clinical trial investigating a vaccine or drug in the four weeks preceding the study.
6. Have received any vaccine in the four weeks preceding the study.
7. Are deprived of freedom by an administrative or court order or in an emergency setting or hospitalized without his/her consent.

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from patients presenting themselves to the emergency departments, outpatient clinic or inpatient wards of the participating sites, and who are diagnosed by laboratory tests to be infected with Dengue. Delegated research staff will screen laboratory-confirmed dengue patients with inclusion/exclusion criteria. Each participant will be given an information sheet and informed consent will obtained from him/her before any study procedures.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2018-07-30 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Concentration of serum A2M, CMA1 and VEGFA will be use to predict whether a dengue patient will develop severe disease as defined by WHO 1997 and WHO 2009 classifications. | 7 days
  Blood will be drawn for measurements of serum concentrations of biomarkers via quantitative enzyme-linked immunosorbent assays (ELISA).

SECONDARY OUTCOMES:
Number of participants develop Dengue Haemorrhagic fever (DHF) within study periods | 7 days
  Patient symptoms will be accessed using WHO 1997 classification for DHF.
Number of participants develop Dengue Shock Syndrome (DSS) within study periods | 7 days
  Patient symptoms will be accessed using WHO 1997 classification for DSS
Number of participants develop Severe Dengue within study periods | 7 days
  Patient symptoms will be accessed using WHO 2009 classification for severe dengue)
Cost of dengue treatments for adoption of such a dengue prognostic technology in hospital | 7 days
  Hospital bills from and outpatient care will be collected to calculate the cost of dengue treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Sophia Archuleta, Principal Investigator — National University Hospital, Singapore
Locations (3):
- Singapore (3):
  - Tan Tock Seng Hospital, Singapore
  - Ng Teng Fong General Hospital, Singapore
  - National University Hospital, Singapore

REFERENCES:
- [Background] Lee LK, Earnest A, Carrasco LR, Thein TL, Gan VC, Lee VJ, Lye DC, Leo YS. Safety and cost savings of reducing adult dengue hospitalization in a tertiary care hospital in Singapore. Trans R Soc Trop Med Hyg. 2013 Jan;107(1):37-42. doi: 10.1093/trstmh/trs009. PMID 23296696
- [Background] Ingram PR, Mahadevan M, Fisher DA. Dengue management: practical and safe hospital-based outpatient care. Trans R Soc Trop Med Hyg. 2009 Feb;103(2):203-5. doi: 10.1016/j.trstmh.2008.07.007. Epub 2008 Aug 29. PMID 18760815
- [Background] Bhatt S, Gething PW, Brady OJ, Messina JP, Farlow AW, Moyes CL, Drake JM, Brownstein JS, Hoen AG, Sankoh O, Myers MF, George DB, Jaenisch T, Wint GR, Simmons CP, Scott TW, Farrar JJ, Hay SI. The global distribution and burden of dengue. Nature. 2013 Apr 25;496(7446):504-7. doi: 10.1038/nature12060. Epub 2013 Apr 7. PMID 23563266
- [Background] Brady OJ, Gething PW, Bhatt S, Messina JP, Brownstein JS, Hoen AG, Moyes CL, Farlow AW, Scott TW, Hay SI. Refining the global spatial limits of dengue virus transmission by evidence-based consensus. PLoS Negl Trop Dis. 2012;6(8):e1760. doi: 10.1371/journal.pntd.0001760. Epub 2012 Aug 7. PMID 22880140
- [Background] Chawla S, Sahoo SS, Singh I, Verma M, Gupta V, Kumari S. Dengue vaccine: come let's fight the menace. Hum Vaccin Immunother. 2015;11(2):474-6. doi: 10.4161/21645515.2014.981077. PMID 25695523